CLINICAL TRIAL: NCT00969280
Title: Acupuncture for Dry Eye Syndrome : A Randomized, Patient-Assessor Blinded, Non-acupuncture Point Shallow Penetration-Controlled Study
Brief Title: Acupuncture for Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Choi, sun-mi/Principal Investigator, Department of Medical Research, Korea Institute of Oriental Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KI0906
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-09

CONDITIONS: Dry Eye Syndromes
Keywords: Acupuncture; Dry eye syndrome; Ocular Surface Disease Index; Schirmer test; Tear film Break-up time
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standardized Acupuncture group (Experimental)
  Interventions: Device: Standardized Acupuncture
- Non-acupoint shallow penetration group (Placebo Comparator)
  Interventions: Device: Non-acupuncture point shallow penetration acupuncture

INTERVENTIONS:
Device: Standardized Acupuncture — Acupuncture treatment will be applied 3 times per week, total 9 times for 3 weeks.
  According to the guideline of WHO standard acupuncture point locations in the western pacific region, acupuncture treatment will be offered in all 17 acupoints: both BL2, GB14, TE23, Extra-1(Taiyang), ST1 and GB 20, and GV23, and Left SP3, LU9, LU10 and HT8, which are located in periorbit, forehead or temple of the head and Lt. forearm and back of the Lt. foot by a disposable 20*30mm (Dongbang Co., korea) acupuncture needle.
  All the acupuncture needles will be inserted, induced strong 'deqi' sensation and retained for 20 minutes.
  Arms: Standardized Acupuncture group
Device: Non-acupuncture point shallow penetration acupuncture — Acupuncture treatment will be applied 3 times per week, all 9 times for 3 weeks.
  Acupuncture treatment will be offered in 17 non-acupuncture points by a disposable 20*30mm acupuncture needle. A strong 'deqi' sensation will not be induced, but inserted acupunctures will be leaved for 20 minutes.
  Arms: Non-acupoint shallow penetration group

SUMMARY:
This study is about the effectiveness of acupuncture treatment on dry eye syndrome. Study hypothesis is that a standardized acupuncture would be more effective than a sham acupuncture in dry eye syndrome patients. This is a randomized, patients-assessor blinded, sham acupuncture controlled study. Additionally, the investigators will assess the safety of acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had dry eye syndromes in single eye or in both eyes e.g. Other disorders of lacrimal gland: Dry eye syndrome (ICD-10: H04.1). He or she must have both of the conditions below:

  1. Patients who have had such symptoms like ocular itching, ocular foreign body sensation, ocular burning, ocular pain, ocular dryness, blurred vision, sensation of photophobia, ocular redness, sensation of tearing
  2. Patient whose tear film break-up time (BUT) is below 10 seconds and measured tear amount is below 10mm/5sec by Schirmer 1 test

Exclusion Criteria:

* Those who have defects of eyelid or eyelashes
* Those who have acute infection of eyelid, eyeball or accessories of eye
* Those who have Stevens-Johnson syndromes or Pemphigoids
* Those who have Vitamin A deficiency
* Those who have any defects of eye or accessories of eye by external injuries
* Those who have undergone any surgical operation for eye during last 3 months
* Those who are using contact lens
* Those who have any difficulties about eye opening or eye closing due to facial palsy
* Those who have undergone punctual occlusion surgery
* Those who have used any kinds of anti-inflammatory eyedrops for recent 2 weeks (steroids, cyclosporin or autologous serum eyedrops)
* Those who have systemic immune therapy
* Those who are pregnant or have any plan for pregnancy
* Those who are not appropriate to this study by investigators decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunmi Choi, doctor, Study Director — Korea Institute of Oriental Medicine; Taehun Kim, Doctor, Principal Investigator — Korea Institute of Oriental Medicine; Mi-suk Shin, Master, Principal Investigator — Korea Institute of Oriental Medicine
Locations (1):
- Clinical Research Center, Korea institute of oriental medicine, Daejeon, Chongchungdo, South Korea

REFERENCES:
- [Derived] Kim TH, Kim JI, Shin MS, Lee MS, Choi JY, Jung SY, Kim AR, Seol JU, Choi SM. Acupuncture for dry eye: a randomised controlled trial protocol. Trials. 2009 Dec 3;10:112. doi: 10.1186/1745-6215-10-112. PMID 19958541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 15 September 2009 to 27 October 2009. Through the advertisements in regional newspapers or university websites, patients were recruited at the clinical research center of the Korea Institute of Oriental Medicine (KIOM) in Daejeon University hospital, Daejeon, Korea.
Pre-assignment Details: 49 participants were tested for eligibility. 6 were excluded because of the insufficient pre-allocation test, denied informed consent and other reasons. After 1 week run-in period, 1 participant was excluded for withdrawal of informed consent. After all, 42 participants were included in this trial.
Groups:
- Standardized Acupuncture Group: Acupuncture treatement was conducted by licensed oriental medicine doctore. total nine acupuncture treatment sessions (three times per week for three weeks)were offered in treatment group. According to Korean traditional theory, 17 acupuncture points were selected for acupuncture (GV23; bilateral BL2, GB14, TE23, Ex1, ST1 and GB20; and unilateral SP3, LU9, LU10 and HT8, on the left for men and right for women), and acupunctures were retained for 20 minutes after "de qi" manipulation for the verum acupuncture group.
- Non-acupoint Shallow Penetration Group: 17 sham points were selected and acupunctures were also retained for 20 minutes after shallow penetration of the skin without any other manipulation for total 9 sessions. The sham points were as follows: both points 2 cm lateral to ST4, 2 cm below ST7, at the parietal eminence of the head, 2 cm internal to ST9, 10 cm internal to BL57, 1.5 cm internal to ST36, single points at the left middle point of the biceps brachii muscle belly, points at 2 cm, 4 cm and 6 cm from the Lt. wrist fold, and one point located between the Lt. 3rd and 4th metatarsophalangeal joints.
Period: Overall Study
Arm/Group | Standardized Acupuncture Group | Non-acupoint Shallow Penetration Group
Started | 21 | 21
Completed | 19 | 18
Not Completed | 2 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — infection of influenza A(H1N1) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standardized Acupuncture Group | Non-acupoint Shallow Penetration Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.52 (11.8) | 42.76 (9.59) | 41.64 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index : OSDI
Description: The OSDI is a questionnaire that consists of 12 questions about ocular irritation and the effect of dry eye on vision. For every question, participants checked at a score between 0 and 4, where 0 equals "none of the time" and 4 equals "all of the time". OSDI scores will be calculated according to the following formula: OSDI = [(sum of scores for all questions answered)*100] / [(total number of questions answered)*4]. The possible range of the OSDI score is 0 to 100. Mean difference of the OSDI scores was calculated from the OSDI scores between Visit 11 and baseline.
Time Frame: Visit 11 (after 3 weeks from baseline)
Population: Statistical analyses were conducted on an intention-to-treat basis (ITT analysis, significance p<0.05). According to the last observation carried forward method (LOCF method), the last observed missing values were used to complete missing values from drop-out participants.
Measure: Mean (Standard Deviation); unit: Scores on the OSDI score
Units Other Than Participants: Eye symptoms
Arm/Group | Standardized Acupuncture Group | Non-acupoint Shallow Penetration Group
Number analyzed (Participants) | 21 | 21
Number analyzed (Eye symptoms) | 21 | 21
Scores on the OSDI score | -17.61 (15.61) | -17.20 (18.81)

2. Secondary Outcome: Visual Analogue Scale of Self Symptoms
Time Frame: every visit
Reporting Status: Not Posted

3. Secondary Outcome: Schirmer 1 Test
Time Frame: visit 1,10
Reporting Status: Not Posted

4. Secondary Outcome: Tear Film Break-up Time : BUT
Time Frame: Visit 1, 10
Reporting Status: Not Posted

5. Secondary Outcome: Medication Quantification Scale (MQS)
Time Frame: every visit
Reporting Status: Not Posted

6. Secondary Outcome: General Assessment
Time Frame: visit 11
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Standardized Acupuncture Group | Non-acupoint Shallow Penetration Group
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No